CLINICAL TRIAL: NCT05799118
Title: Study of the Role of Genetic Modifiers in Hemoglobinopathies
Acronym: INHERENT
Status: Recruiting | Type: Observational
Sponsor: Cyprus Institute of Neurology and Genetics (Other)
Responsible Party: Principal Investigator, Petros Kountouris, PhD, Associate Scientist, Lead of the Biomedical and Translational Informatics Group, Molecular Genetics Thalassaemia Department, Cyprus Institute of Neurology and Genetics
Other Study IDs: 1
Record Dates: First submitted 2023-03-10; First posted 2023-04-05 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Sickle Cell Disease; Thalassemia, Beta; Thalassemia Alpha; Hemoglobinopathies
Keywords: GWAS; thalassemia; sickle cell disease; genetic modifiers
MeSH Terms: conditions — Anemia, Sickle Cell; beta-Thalassemia; alpha-Thalassemia; Hemoglobinopathies; Thalassemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort: Individuals with hemoglobinopathies
  Interventions: Genetic: GWAS

INTERVENTIONS:
Genetic: GWAS — The study will perform a GWAS experiments for all recruited subjects. The blood sample will be collected during routine clinical visits, only if DNA is not already available in existing biobanks. All individuals will provide consent for participation in the study.

SUMMARY:
This study will investigate the role of genetic modifiers in hemoglobinopathies through a large-scale, multi-ethnic genome-wide association study (GWAS).

DETAILED DESCRIPTION:
Hemoglobinopathies, including sickle cell disease (SCD) and beta-thalassemia, are prevalent diseases with variable clinical manifestation and severity that are thought to be governed, in part, by genetic modifiers. Despite the identification and characterization of a few putative genetic modifiers by previous studies, these are as yet insufficient to guide treatment recommendations or risk-stratify patients reliably. Also, it is expected that many additional genetic variants exist that can modify disease and its severity. This large-scale genome-wide association study (GWAS) will utilize SNP chips to investigate the genetic profile of individuals with hemoglobinopathies, thereby addressing the challenges of previous studies related to small sample sizes and low statistical power, while promoting the participation of diverse populations worldwide. The study aims to i) discover new genetic modifiers of hemoglobinopathies, ii) validate previously reported genetic modifiers, iii) pool and analyze existing genomic data, iv) standardize phenotypic descriptions, v) develop a research resource of disease-specific data generated in INHERENT, including genomic, phenotypic, and functional data, and vi) develop risk scores that can be used for patient stratification.

The main endpoints include:

1. Worldwide demography, including numbers of patients, main genotypes, and overall disease severity/burden in participating centres
2. Genetic modifiers affecting clinical or laboratory phenotypes of hemoglobinopathies, including

   1. overall survival in SCD and/or thalassemia,
   2. stroke and/or decreased neurocognitive function in SCD and/or thalassemia,
   3. renal impairment in SCD and/or thalassemia,
   4. leg ulcers in SCD,
   5. priapism in SCD,
   6. mild or severe acute pain and/or chronic pain syndromes in SCD,
   7. pulmonary hypertension in SCD and/or thalassemia,
   8. hyperhemolysis in SCD and/or thalassemia,
   9. fetal hemoglobin levels,
   10. degree of ineffective erythropoiesis,
   11. hepatic fibrosis/cirrhosis and/or cardiac siderosis,
3. Genetic modifiers affecting response to treatment, including

   1. response to hydroxyurea,
   2. response to iron chelation treatment,
   3. response to emerging therapeutic agents

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of an inherited hemoglobinopathy, including sickle cell disease (SCD), β-thalassemia, and α-thalassemia; all genotypes will be considered.
* Age ≥ 2 years old at the time of the collection of the phenotypic data.
* There will be no limits on study participants in terms of gender, ethnicity, morbidities.

Exclusion Criteria:

* Patients treated with stem cell transplantation or genetic therapy.
* Age < 2 years old at the time of the collection of the phenotypic data.
* Patient or legal representative for minors unwilling or unable to give consent.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals diagnosed with an inherited hemoglobinopathy and are under regular follow-up in the participating centers
Sampling Method: Non-Probability Sample
Enrollment: 30000 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Genetic modifiers in haemoglobinopathies through GWAS | 5 years
  Number of genetic variants (SNPs) associated with disease-specific phenotypes

CONTACTS AND LOCATIONS:
Overall Officials: Petros Kountouris, PhD, Principal Investigator — Cyprus Institute of Neurology and Genetics
Locations (26):
- Boston Children's Hospital, Boston, Massachusetts, United States
- Lucrecia Paím Maternity, Luanda, Angola
- University of Buenos Aires, Buenos Aires, Argentina
- University Hospitals Leuven, Leuven, Belgium
- Universiti Brunei Darussalam, Brunei, Brunei
- Cyprus (4):
  - Larnaca General Hospital, Larnaca
  - Limassol General Hospital, Limassol
  - Archbishop Makarios III Hospital, Nicosia
  - Paphos General Hospital, Paphos
- Centre Hospitalier Monkole, Kinshasa, Democratic Republic of the Congo
- Rigshospitalet, Copenhagen, Denmark
- Greece (4):
  - Hippokrateio Hospital of Athens, Athens
  - Laiko General Hospital, Athens
  - National and Kapodistrian University of Athens, Athens
  - General Hospital of Larissa, Larissa
- Emek Medical Centre, Afula, Israel
- University of Turin, Turin, Italy
- Malaysia (3):
  - Ampang Hospital, Ampang
  - Universiti Kebangsaan Malaysia, Bangi
  - Universiti Sains Malaysia, Kota Bharu
- Nigeria (3):
  - University of Abuja, Abuja
  - Kaduna State University, Kaduna
  - Ahmadu Bello University, Zaria
- University of Lahore, Lahore, Pakistan
- Centro Hospitalar e Universitário de Coimbra, Coimbra, Portugal
- Hospital Clínico San Carlos, Madrid, Spain

REFERENCES:
- [Background] Kountouris P, Stephanou C, Archer N, Bonifazi F, Giannuzzi V, Kuo KHM, Maggio A, Makani J, Manu-Pereira MDM, Michailidou K, Nkya S, Nnodu OE, Trompeter S, Tshilolo L, Wonkam A, Zilfalil BA, Inusa BPD, Kleanthous M; on behalf of the International Hemoglobinopathy Research Network (INHERENT). The International Hemoglobinopathy Research Network (INHERENT): An international initiative to study the role of genetic modifiers in hemoglobinopathies. Am J Hematol. 2021 Nov 1;96(11):E416-E420. doi: 10.1002/ajh.26323. Epub 2021 Aug 30. No abstract available. PMID 34406671
- See also: Official INHERENT website — https://inherentnetwork.org